CLINICAL TRIAL: NCT01036308
Title: Comparison of the Effects of Three Native Legume Kernel Fibres on Cholesterol Metabolism in Healthy Subjects
Brief Title: Intervention With Legume Kernel Fibre in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Prof. Dr. G. Jahreis, Friedrich Schiller University Jena, Department of Nutritional Physiology
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LSEP H32-07
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2009-12

CONDITIONS: Healthy
Keywords: dietary fibre; legumes; lupin kernel fibre; soy fibre; bile acids; short-chain fatty acids; cholesterol metabolism; Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TypTop (Experimental): Lupinus albus Typ Top (lupin kernel fibre, dietary fibre content: 83%)
  Interventions: Dietary Supplement: pure fibre-product; Dietary Supplement: reference fibre
- Soy fibre (Experimental): Glycine max Hefeng (soy fibre; dietary fibre content: 77%)
  Interventions: Dietary Supplement: pure fibre-product; Dietary Supplement: reference fibre
- Boregine (Experimental): Lupinus angustifolius Boregine (lupin kernel fibre, dietary fibre content: 87%)
  Interventions: Dietary Supplement: pure fibre-product; Dietary Supplement: reference fibre

INTERVENTIONS:
Dietary Supplement: pure fibre-product — The subjects consumed 25 g pure fibre-product per day over two weeks. One half a portion of the fibres was stirred into a selected milk product and the other half in juice.
Dietary Supplement: reference fibre — The subjects consumed 25 g reference fibre (citrus fibre: Herbacel AQ Plus; Herbafood Ingredients) per day over two weeks. One half a portion of the fibres was stirred into a selected milk product and the other half in juice.
  Other Names: Herbacel AQ Plus; citrus fibre

SUMMARY:
The objective of the conducted study was to determine the efficacy of the native legume kernel fibres of Lupinus angustifolius Boregine (Boregine), Lupinus albus Typ Top (TypTop) and Glycine max Hefeng (Soy fibre) on prevention of risk factors for gastrointestinal or cardiovascular diseases.

DETAILED DESCRIPTION:
Dietary fibre is suspected to effect the faecal concentration and excretion of bile acids by binding the bile acids and by increasing the faecal mass. Bile acids, especially the secondary bile acids, are potential risk factors for colorectal cancer. A high bile acid-binding ability of fibre could lead to lower serum cholesterol concentrations by interrupting the enterohepatic circulation. There is evidence that the consumption of legume kernel fibre, containing both soluble and insoluble fibre fractions, may beneficially modify bowel health.

Seventy-eight healthy volunteers were enrolled. Seventy-six subjects (mean age of 24 years, 55 women and 21 men) completed the double-blind, randomized crossover trial. After two weeks run-in period, half of the volunteers consumed 25 g of legume fibres (Boregine, TypTop or Soy fibre) every day, and the other half received a reference fibre product (citrus fibre, Herbacel AQ Plus) for a period of two weeks. After two weeks wash-out the intervention changed between the groups.

At the end of each period a quantitative stool and urine collection took place and fasting blood samples were drawn.

ELIGIBILITY:
Inclusion Criteria:

* age 20-45 years
* healthy subjects

Exclusion Criteria:

* intake of pharmaceuticals and nutritional supplements
* allergy against legumes
* intolerance against milk protein
* pregnancy, lactation
* chronic diseases

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2007-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Changes of serum lipids (cholesterol metabolism) | after 2, 4 and 8 weeks

SECONDARY OUTCOMES:
Changes of general excretion parameters, neutral sterols, bile acids, short-chain fatty acids, fibre excretion | after 2, 4 and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Jahreis, Prof. Dr., Principal Investigator — Friedrich Schiller University Jena, Institute of Nutrition, Department of Nutrional Physiology
Locations (1):
- Friedrich Schiller University Jena, Institute of Nutrition, Department of Nutrional Physiology, Jena, Thuringia, Germany

REFERENCES:
- [Derived] Fechner A, Fenske K, Jahreis G. Effects of legume kernel fibres and citrus fibre on putative risk factors for colorectal cancer: a randomised, double-blind, crossover human intervention trial. Nutr J. 2013 Jul 16;12:101. doi: 10.1186/1475-2891-12-101. PMID 24060277